CLINICAL TRIAL: NCT01249898
Title: The Treatment and Intra-operative Imaging of Scaphoid Fracture Reduction and Fixation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Shai Luria, Hadassah Medical Organization
Other Study IDs: Luria004-HMO-CTIL
Record Dates: First submitted 2010-11-28; First posted 2010-11-30 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Scaphoid Fractures
Keywords: Fracture in the Scaphoid fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Scaphoid fractures are the most common carpal bone fractures, and second most common wrist fractures (second to distal radius fractures). Lack of proper immobilization or displacement of these fractures commonly results in fracture nonunion or malunion followed by the development of wrist post-traumatic osteoarthritis. In addition, proper reduction and fixation of these fractures are challenging to the most experienced hand surgeons.

The investigators are going to follow-up the patients population suffering from Scaphoid fractures(nonunion included) for one year. The investigators will evaluate this follow up results in two ways:

1. Intra-operative imaging of scaphoid fracture fixation - feasibility evaluation.
2. Treatment of scaphoid fracture non-union.

ELIGIBILITY:
Inclusion Criteria:

1. Ages of 18 and 60 during the study period;
2. Scaphoid fractures to be operatively reduced and fixated, including fracture non-unions;
3. Signed informed consent.

Exclusion Criteria:

1. Non-displaced fractures of the scaphoid.
2. Soldiers in active military service.
3. pregnant women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that suffer fron Scaphoid fractures(nonunion included).
Sampling Method: Probability Sample

PRIMARY OUTCOMES:
Intra-operative imaging of scaphoid fracture fixation - feasibility evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organizaton, Jerusalem, Israel